CLINICAL TRIAL: NCT06561269
Title: Ultrasound_guided Multifidus Plane Block Versus Ultrasound_guided Caudal Block for Pediatric Hypospadias Surgery: a Randomized Controlled Clinical Trial
Brief Title: Multifidus Plane Block Versus Caudal Block for Hypospadias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Tarek, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD73/2024
Record Dates: First submitted 2024-06-02; First posted 2024-08-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-04

CONDITIONS: Hypospadias; Caudal Block
Keywords: Hypospadias; caudal block
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifidus plane block (MPB) group (Experimental): Participants will be injected bupivacaine at the fascial plane between the multifidus muscle and the median sacral crests of S2 and S3
  Interventions: Procedure: Multifidus plane block
- Caudal block (CB) group (Experimental): Participants will be injected by bupivacaine, between the two sacral cornua
  Interventions: Procedure: caudal block

INTERVENTIONS:
Procedure: Multifidus plane block — Using the "in-plane" technique,The fascial plane between the multifidus muscle and the median sacral crests of S2 and S3, will be injected by bupivacaine.
  Arms: Multifidus plane block (MPB) group
Procedure: caudal block — The ultrasound transducer will first be placed transversely at the midline to obtain the transverse view of sacral hiatus. At this level, the ultrasound transducer is rotated 90 degrees to obtain the longitudinal view of sacral hiatus. The block needle is inserted using the "in-plane" technique.
  Arms: Caudal block (CB) group

SUMMARY:
This study aims to evaluate the safety and efficacy of ultrasound-guided sacral multifidus plane block and compare its analgesic effect to ultrasound-guided caudal block in pediatric patients undergoing hypospadias surgery under general anesthesia

DETAILED DESCRIPTION:
Peri-operative pain management in pediatric surgeries is considered a challenging issue for the anesthesiologists. The usage of regional anesthesia in association with general anesthesia (GA) is a simple intraoperative way that reduces (GA) requirements and side effects. Recently, paraspinal fascial plane block, the sacral multifidus plane block (MPB), was used successfully in infants. The study has been designed to determine the effect of MPB versus caudal epidural block to control peri-operative pain in hypospadias surgeries in children.

ELIGIBILITY:
Inclusion Criteria:

* ⦁ Children aged (1 -7) years old.

  * All patients will be of ASA classification I, II physical status

Exclusion Criteria:

* ⦁ Parents refusing to participate are excluded from the trial.

  * Children who had spinal anomalies, altered mental status.
  * A history of developmental delay.
  * Blood diseases: Coagulopathy or anaemia.
  * Infection at the site of injection.
  * Drug allergy.

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Children aged (1 -7) years old.All patients will be of ASA classification I, II physical status
Enrollment: 30 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
is to measure the first time to rescue analgesia postoperative (24 hours). | 24 hours postoperative
  Measure the first time to rescue analgesia post operative

SECONDARY OUTCOMES:
Heart rate | start to end of surgery
  measuring HR changes
Blood pressure | start to end of the surgery.
  measuring BP changes

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt